CLINICAL TRIAL: NCT03398915
Title: The European Robotic Spinal Instrumentation (EUROSPIN) Study: A European Prospective Multicenter Multinational Pragmatic Trial on Robot-guided Versus Navigated Versus Freehand Pedicle Screw Fixation
Brief Title: The European Robotic Spinal Instrumentation (EUROSPIN) Study
Acronym: EUROSPIN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Marc Schröder (Other)
Responsible Party: Sponsor-Investigator, Marc Schröder, Head of Department, Bergman Clinics
Organization: Bergman Clinics (Other)
Other Study IDs: EUROSPIN
Record Dates: First submitted 2018-01-07; First posted 2018-01-16 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Degenerative Disc Disease; Spondylolisthesis; Spinal Stenosis; Recurrent Disc Herniation; Spondylodiskitis; Spinal Tumor; Spinal Metastases
Keywords: robotic; robot-guided; navigated; computer-assisted; pedicle screw; instrumentation; thoracolumbar
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spondylolisthesis; Spinal Stenosis; Intervertebral Disc Displacement; Discitis; Spinal Cord Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Robot-Guided Transpedicular Instrumentation: This arm will comprise all patients that receive transpedicular instrumentation by use of a robotic guidance system (SpineAssist or Renaissance, Mazor Robotics, Ltd., Caesarea, Israel or ROSA Spine, Medtech, Montpellier, France).
  Interventions: Procedure: Transpedicular Instrumentation
- Navigated Transpedicular Instrumentation: This arm will comprise all patients that receive transpedicular instrumentation by use of navigation (computer assistance using CT, O-arm or 3D-fluoroscopic imaging).
  Interventions: Procedure: Transpedicular Instrumentation
- Freehand Transpedicular Instrumentation: This arm will comprise all patients that receive transpedicular instrumentation by use of the conventional freehand technique.
  Interventions: Procedure: Transpedicular Instrumentation

INTERVENTIONS:
Procedure: Transpedicular Instrumentation — Transpedicular screw placement and instrumentation

SUMMARY:
In a multinational prospective study, preoperative, intraoperative, perioperative and follow-up data on patients receiving thoracolumbar pedicle screw placement for degenerative disease or infections or tumors will be collected. The three arms consist of robot-guided (RG), navigated (NV), or freehand (FH) screw insertion.

DETAILED DESCRIPTION:
Introduction A decade ago, minimally invasive surgery (MIS) was considered a promising development in spine surgery, yet the value of the pioneering technologies was questionable. With the growing number of experienced MIS surgeons, the influx of evidence in favour of MIS is rapidly increasing. This makes a compelling argument towards MIS offering distinct clinical benefits over open approaches in terms of blood loss, length of stay, rehabilitation, cost-effectiveness and perioperative patient comfort. Due to the limited or inexistent line-of-sight in MIS procedures, surgeons need to rely on imaging, navigation, and guidance technologies to operate in a safe and efficient manner. Therefore, a plethora of new and ever improving navigational systems have been developed. These systems allow a consistent level of safety and accuracy, on par with results achieved by very experienced free hand surgeons, with a reasonably short learning curve. Computer-based navigation systems were first introduced to spine surgery in 1995 and while they have been long established as standards in certain cranial procedures, they have not been similarly adopted in spine surgery.

Designed to overcome some of the limitations of navigation-based technologies, robot-guided surgery has become commercially available to surgeons worldwide, like SpineAssist® (Mazor Robotics Ltd. Caesarea, Israel) and the recently launched ROSA™ Spine (Zimmer-Biomet, Warsaw, Indiana, USA). These systems are rapidly challenging the gold standards. SpineAssist®, and its upgraded version, the Renaissance®, provides a stable drilling platform and restricts the surgeon's natural full range of motion to 2 degrees of freedom (up/down motion and yaw in the cannula). The system's guidance unit moves into the trajectory based on exact preoperative planning of pedicle screws, while accounting for changes in intervertebral relationships such as due to distraction, cage insertion or changes between the supine patient position in the preoperative CT and the prone patient on the operating table. Published evidence on robot-guided screw placement has demonstrated high levels of accuracy with most reports ranging around 98% of screws placed within the pedicle or with a cortical encroachment of less than 2 mm.4 Although the reliability and accuracy of robot-guided spine surgery have been established, the actual benefits for the patient in terms of clinical outcomes and revision surgeries remain unknown. We have recently conducted cohort studies that showed some evidence that robotic guidance lowers the rate of intraoperative screw revisions and implant related reoperations compared to free hand procedures, while achieving comparable clinical outcomes. We now want to assess these factors, among others, on a higher level of evidence. We aim to conduct a prospective, multicenter, multinational controlled trial comparing clinical and patient reported outcomes of robotic guided (RG) pedicle screw placement vs. navigated (NV) vs. free hand (FH) pedicle screw placement using pooled data from three centers.

Study Design The European Robotic Spinal Instrumentation (EUROSPIN) study is a prospective, international, multicentre, pragmatic, open-label, non-randomized controlled trial comparing the effectiveness of three techniques for pedicle screw instrumentation, namely RG, NV (CT-, O-Arm, or 3DFL-based), and FH. Following the baseline evaluation, patients will receive one of the three treatments, and will subsequently be followed up for 24 months (Figure 1). The primary analysis will be conducted using the 12-month data.

Sample Size Calculation It was determined that, to detect an intergroup difference of 5% in the primary endpoint, 205 patients are required per group to achieve a power of 1 - beta = 0.8 at alpha = 0.05. The incidence rates were based on the published literature, with an approximated incidence rate of the primary endpoint of 0% for the intervention and 5% for the control group. Because the study protocol is in line with the normal clinical follow-up of most centers, a low dropout rate is expected. This led to a minimum total sample size of 615 patients.

Monitoring An epidemiologist from the sponsor institution will organize an initiation monitor visit at every participating center before starting recruitment. This monitor visit will check whether all study staff are properly trained and the delegation of tasks are well documented (complete Investigator Site File, training and delegation logs). An additional audit will be carried out at 6 months after initiation of recruitment to check whether source documentation and eCRF documentation is similar. Throughout the entire study additional queries by the monitor are send to the investigator in the data capturing system to ensure proper data capturing.

ELIGIBILITY:
Inclusion Criteria

* Informed consent
* Thoracolumbar pedicle screw placement
* Indication for surgery: Degenerative pathologies (stenosis, spondylolisthesis, degenerative disc disease, recurrent disc herniation), infections, tumors, fractures, trauma
* Age ≥ 18

Exclusion Criteria

* Deformity surgery
* >5 index levels

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving thoracolumbar transpedicular screw placement for degenerative pathologies (stenosis, spondylolisthesis, degenerative disc disease, recurrent disc herniation), infections, fractures, trauma, or tumors.
Sampling Method: Non-Probability Sample
Enrollment: 615 (Estimated)
Dates: Start 2018-02-20 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Revision surgery for a malpositioned pedicle screw | 12 months
  We defined the primary endpoint as required revision surgery for a malpositioned or loosened pedicle screw within the first postoperative year.

SECONDARY OUTCOMES:
Intraoperative screw revision | Intraoperative
  Revision or redirection of a placed screw during the same general anesthesia session
Duration of Surgery | Intraoperative
  Duration of Surgery in minutes
Length of Hospital Stay | Through hospital stay (From admission to discharge of the hospital stay in which the primary surgery was carried out)
  Length of Hospital Stay in days (Defined as from admission to discharge, during the hospital stay in which the primary surgery was carried out)
Radiation Dose (DAP) | Intraoperative
  Radiation Dose as DAP (Dose Area Product, cGy cm2)
Estimated Blood Loss | Intraoperative
  Estimated Blood Loss (ml)
Need for blood transfusion | Through hospital stay (From admission to discharge of the hospital stay in which the primary surgery was carried out)
  Need for blood transfusion during the hospital stay (Defined as from admission to discharge, during the hospital stay in which the primary surgery was carried out)
Intraoperative Complications | 0 weeks
  Intraoperative Complications
Postoperative Complications | 6 weeks
  Postoperative Complications
EQ-5D-3L | 2 years
  EQ-5D-3L (Health-related quality of life) EuroQOL-five dimensions 3-level version measures health-related quality of life.
  The scale is subdivided into an index, ranging from 0 to 1 and normalized to population-specific values, and a "thermometer" or visual analogue scale, ranging from 0 to 100.
  The two subscores are not combined towards a single score. Higher values represent a better health-related quality of life in both subscores.
NRS back pain severity | 2 years
  Numeric Rating Scale (NRS) of back pain severity The scale ranges from 0 to 10. Only integers are available to choose from. Higher values represent a higher amount of pain. There are no subscales.
NRS leg pain severity | 2 years
  Numeric Rating Scale (NRS) of leg pain severity The scale ranges from 0 to 10. Only integers are available to choose from. Higher values represent a higher amount of pain. There are no subscales.
Oswestry Disability Index | 2 years
  Oswestry Disability Index (ODI) for functional impairment

OTHER OUTCOMES:
Frequency of use of analgetics | 2 years
  Frequency of use of analgetics (daily/weekly/not regularly)
Satisfaction with symptoms | 2 years
  Satisfaction with symptoms (satisfied/neutral/dissatisfied)
Smoking status | 2 years
  Smoking status (active/ceased/never)
Working status | 2 years
  Working status (able to work/unable to work)
Return to work | 2 years
  Return to work (number of weeks/not yet)
Overall rate of reoperations | 2 weeks
  Overall rate of reoperations

CONTACTS AND LOCATIONS:
Overall Officials: Victor E Staartjes, BMed, Study Director — Department of Neurosurgery, Bergman Clinics; Marc L Schröder, MD, PhD, Principal Investigator — Department of Neurosurgery, Bergman Clinics; Paulien M van Kampen, PhD, Study Director — Department of Epidemiology, Bergman Clinics
Locations (13):
- Medical University of Innsbruck, Innsbruck, Austria
- France (2):
  - Amiens University Hospital, Amiens
  - La Pitié Salpetrière Hospital, Paris
- Germany (5):
  - HELIOS Klinikum Berlin-Buch, Berlin
  - Ortho-Klinik Dortmund, Dortmund
  - Universitätsmedizin Göttingen, Göttingen
  - Klinikum Rechts der Isar, Munich
  - St Josef Brothers Hospital, Paderborn
- Netherlands (3):
  - Martini Hospital, Groningen
  - Bergman Clinics, Naarden
  - MC Haaglanden, The Hague
- Switzerland (2):
  - HUG Geneva, Geneva
  - Clinique de La Source, Lausanne

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Goldstein CL, Phillips FM, Rampersaud YR. Comparative Effectiveness and Economic Evaluations of Open Versus Minimally Invasive Posterior or Transforaminal Lumbar Interbody Fusion: A Systematic Review. Spine (Phila Pa 1976). 2016 Apr;41 Suppl 8:S74-89. doi: 10.1097/BRS.0000000000001462. PMID 26825793
- [Background] Hu X, Lieberman IH. What is the learning curve for robotic-assisted pedicle screw placement in spine surgery? Clin Orthop Relat Res. 2014 Jun;472(6):1839-44. doi: 10.1007/s11999-013-3291-1. PMID 24048889
- [Background] Schatlo B, Martinez R, Alaid A, von Eckardstein K, Akhavan-Sigari R, Hahn A, Stockhammer F, Rohde V. Unskilled unawareness and the learning curve in robotic spine surgery. Acta Neurochir (Wien). 2015 Oct;157(10):1819-23; discussion 1823. doi: 10.1007/s00701-015-2535-0. Epub 2015 Aug 19. PMID 26287268
- [Background] Marcus HJ, Cundy TP, Nandi D, Yang GZ, Darzi A. Robot-assisted and fluoroscopy-guided pedicle screw placement: a systematic review. Eur Spine J. 2014 Feb;23(2):291-7. doi: 10.1007/s00586-013-2879-1. Epub 2013 Jun 26. PMID 23801017
- [Background] Schroder ML, Staartjes VE. Revisions for screw malposition and clinical outcomes after robot-guided lumbar fusion for spondylolisthesis. Neurosurg Focus. 2017 May;42(5):E12. doi: 10.3171/2017.3.FOCUS16534. PMID 28463610
- [Background] Molliqaj G, Schatlo B, Alaid A, Solomiichuk V, Rohde V, Schaller K, Tessitore E. Accuracy of robot-guided versus freehand fluoroscopy-assisted pedicle screw insertion in thoracolumbar spinal surgery. Neurosurg Focus. 2017 May;42(5):E14. doi: 10.3171/2017.3.FOCUS179. PMID 28463623
- [Background] Schatlo B, Molliqaj G, Cuvinciuc V, Kotowski M, Schaller K, Tessitore E. Safety and accuracy of robot-assisted versus fluoroscopy-guided pedicle screw insertion for degenerative diseases of the lumbar spine: a matched cohort comparison. J Neurosurg Spine. 2014 Jun;20(6):636-43. doi: 10.3171/2014.3.SPINE13714. Epub 2014 Apr 11. PMID 24725180
- [Background] Rabin R, de Charro F. EQ-5D: a measure of health status from the EuroQol Group. Ann Med. 2001 Jul;33(5):337-43. doi: 10.3109/07853890109002087. PMID 11491192
- [Background] Fairbank JC, Couper J, Davies JB, O'Brien JP. The Oswestry low back pain disability questionnaire. Physiotherapy. 1980 Aug;66(8):271-3. No abstract available. PMID 6450426
- [Background] Roland M, Morris R. A study of the natural history of back pain. Part I: development of a reliable and sensitive measure of disability in low-back pain. Spine (Phila Pa 1976). 1983 Mar;8(2):141-4. doi: 10.1097/00007632-198303000-00004. No abstract available. PMID 6222486
- [Background] Ostelo RW, Deyo RA, Stratford P, Waddell G, Croft P, Von Korff M, Bouter LM, de Vet HC. Interpreting change scores for pain and functional status in low back pain: towards international consensus regarding minimal important change. Spine (Phila Pa 1976). 2008 Jan 1;33(1):90-4. doi: 10.1097/BRS.0b013e31815e3a10. PMID 18165753
- [Background] R Core Team. R: A Language and Environment for Statistical Computing. (R Foundation for Statistical Computing, 2017).
- [Background] Staartjes VE, Klukowska AM, Schroder ML. Pedicle Screw Revision in Robot-Guided, Navigated, and Freehand Thoracolumbar Instrumentation: A Systematic Review and Meta-Analysis. World Neurosurg. 2018 Aug;116:433-443.e8. doi: 10.1016/j.wneu.2018.05.159. Epub 2018 May 31. PMID 29859354
- [Derived] Staartjes VE, Molliqaj G, van Kampen PM, Eversdijk HAJ, Amelot A, Bettag C, Wolfs JFC, Urbanski S, Hedayat F, Schneekloth CG, Abu Saris M, Lefranc M, Peltier J, Boscherini D, Fiss I, Schatlo B, Rohde V, Ryang YM, Krieg SM, Meyer B, Kogl N, Girod PP, Thome C, Twisk JWR, Tessitore E, Schroder ML. The European Robotic Spinal Instrumentation (EUROSPIN) study: protocol for a multicentre prospective observational study of pedicle screw revision surgery after robot-guided, navigated and freehand thoracolumbar spinal fusion. BMJ Open. 2019 Sep 8;9(9):e030389. doi: 10.1136/bmjopen-2019-030389. PMID 31501123